CLINICAL TRIAL: NCT03395730
Title: Intraumbilical Oxytocin Compared to Placental Cord Drainage in the Management of Third Stage of Labor: A Randomized Controlled Study
Brief Title: Intraumbilical Oxytocin Versus Placental Cord Drainage in the Management of 3rd Stage of Labor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eslam Mohammed Abbas (Other)
Responsible Party: Sponsor-Investigator, Eslam Mohammed Abbas, physician, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ppsi
Record Dates: First submitted 2017-12-28; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Postpartum Haemorrhage With Retained Placenta

STUDY DESIGN:
Intervention Model Description: The present study will be conducted on 150 women recruited from the delivery ward of our hospital after they had received information on the purpose and course of the study from the medical investigator and had provided the written consent during routine prenatal visits , they will be randomly divided into:
  * Group (A) "Study Group 1": (n = 50)
  * Group (B) "Study Group 2": (n = 50)
  * Group (C) "Control Group": (n = 50)
Who Masked: Participant, Care Provider
Masking Description: Randomization will be based on the sequence generation created by computer and the randomization tables will be kept with the study supervisor. Consenting patients fulfilling inclusion criteria will be randomized into one of the following 3 groups. Randomized allocation will be kept in opaque sealed envelopes, with enrollment numbers written on the envelopes. The envelopes will contain a card on with the designated study group will be written. After enrollment of the patients in the study, the envelopes marked with study number will be unsealed and the patients allocated to either groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- • Group (A) "Study Group 1": (Experimental): In the labor room women in Group A (n = 50):
  * Clamping and cutting the placental cord after delivery of the baby.
  * Immediate intraumbilical vein injection of Oxytocin (Syntocinon®) 20 units diluted in 20 ml of 0.9% saline solution
  Interventions: Drug: Intraumbilical vein injection oxytocin
- • Group (B) "Study Group 2": (Experimental): In the labor room women in Group B (n = 50):
  * Clamping and cutting the placental cord after delivery of the baby.
  * Immediate unclamping of the maternal side, allowing the blood to drain freely for a duration of three minutes.
  Interventions: Procedure: placental cord drainage
- • Group (C) "Control Group": (Active Comparator): In the labor room women in Group C (n = 50):
  * Clamping and cutting the placental cord after 2 minutes of delivery of the baby.
  * Placenta will be delivered spontaneously after appearance of clinical signs of placental separation
  Interventions: Procedure: Expectant managment of 3rd stage of labour

INTERVENTIONS:
Drug: Intraumbilical vein injection oxytocin — intraumbilical vein injection of oxytocin 20 units diluted in 20 ml of 0.9% saline solution immediately after delivery of the baby, clamping and cutting the cord.
  Arms: • Group (A) "Study Group 1":
Procedure: placental cord drainage — placental cor drainage immediately after delivery. This scenario will include placental cord clamping and cutting after delivery of the baby followed by immediately unclamping of the maternal side, allowing the blood to drain freely for a duration of three minutes.
  Arms: • Group (B) "Study Group 2":
Procedure: Expectant managment of 3rd stage of labour — Placenta will be delivered spontaneously after appearance of clinical signs of placental separation, which include strong uterine contraction, vaginal bleeding, and descending of umbilical cord through the vulva. This scenario will include placental cord clamping and cutting after 2 minutes of delivery of the baby.
  Arms: • Group (C) "Control Group":

SUMMARY:
The aim of this study is to compare the effectiveness of intraumbilical oxytocin and placental cord drainage in the management of third stage of labor.

Does the use of intraumbilical vein oxytocin injection or the use of Placental cord drainage can cause a reduction of blood loss, Hb level drop, the length of the third stage of labor and the incidence of manual removal of the retained placenta during the third stage of labor in pregnant women after delivery of the infant?

DETAILED DESCRIPTION:
Study:

Study Design: A prospective randomized clinical trial. Study setting: The study will be conducted in Ain Shams University Maternity Hospital.

All pregnant women in the delivery ward will be submitted to:

1. Detailed complete history taking with special emphasis to maternal age, Parity, Maternal weight, as well as presence of any disease.
2. Clinical Examination:

   a. General examination. b. Abdominal examination (Symphysis-fundal height) and pelvic examination.
3. Investigation

   1. Ultrasound assessment to evaluate GA, fetal weight, AFI and Placental site.
   2. Basal complete blood picture, urine analysis and random blood sugar.

      The selected patients will fulfill the following criteria:

      • Pregnant women between 18-35 years of age with normal pregnancy.

      • A singleton fetus at a gestational age of 37 - 42 weeks in a cephalic presentation.

      • Neonatal birth weight of 2500 to 4500 grams.

      Exclusion criteria:

      • Medical disorders and hypertensive disorders of pregnancy.

      • Intrauterine fetal death.

      • Known or suspected fetal anomalies.

      • Oxytocin induction or Augmented cases.
      * Obstetrical complications (bleeding, premature rupture of membranes).
      * Previous CS or Previous Myomectomy.

      Study population:

      The present study will be conducted on 150 women recruited from the delivery ward of our hospital after they had received information on the purpose and course of the study from the medical investigator and had provided the written consent during routine prenatal visits , The 150 study participants will be divided into three groups using simple random distribution technique. After monitoring the duration of active phase and second stage of labor by following the partograph.

      Randomization and Allocation concealment:

      Randomization will be based on the sequence generation created by computer and the randomization tables will be kept with the study supervisor. Consenting patients fulfilling inclusion criteria will be randomized into one of the following 3 groups. Randomized allocation will be kept in opaque sealed envelopes, with enrollment numbers written on the envelopes. The envelopes will contain a card on with the designated study group will be written. After enrollment of the patients in the study, the envelopes marked with study number will be unsealed and the patients allocated to either groups:

      • Group (A) "Study Group 1": In the labor room women in Group A (n = 50) receive intraumbilical vein injection oxytocin 20 units diluted in 20 ml of 0.9% saline solution immediately after delivery of the baby, clamping and cutting the cord.

      • Group (B) "Study Group 2": The women in Group B (n = 50) have placental drainage immediately after delivery. This scenario will include placental cord clamping and cutting after delivery of the baby followed by immediately unclamping of the maternal side, allowing the blood to drain freely for a duration of three minutes.

      • Group (C) "Control Group": The women in Group C (n = 50) as a control group receive no intervention. Placenta will be delivered spontaneously after appearance of clinical signs of placental separation, which include strong uterine contraction, vaginal bleeding, and descending of umbilical cord through the vulva. This scenario will include placental cord clamping and cutting after 2 minutes of delivery of the baby.

      Outcome:

      Retained placenta is defined as a placenta that remained in the uterus for 30 minutes or more after delivery (Begley et al., 2014).
      * 1ry outcome: Duration of the third stage of labor.
      * 2ry outcome: Retained placenta, need for manual removal of placenta and the drop in Hb will be recorded.

      Sample size calculation:

      Sample size was calculated using PASS® version 11 program, sample size calculation was based on study carried out by (Güngördük et al., 2011). A preliminary power analysis was carried out to calculate the sample size using a formula: d = Δ/SD, where d is standardized difference, Δ is the smallest clinically significant difference and SD is standard deviation of the test group. Duration of 1.6 minutes was considered as the smallest clinically significant difference, and the SD (1.6 minutes) was selected the study performed by (Güngördük et al., 2011). Also, a standardized difference of 1.0 was obtained using nomogram. The power analysis suggested that a sample of 50 women in each group would provide a power of 95%, at 5% significance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18-35 years of age with normal pregnancy.
* A singleton fetus at a gestational age of 37 - 42 weeks in a cephalic presentation.
* Neonatal birth weight of 2500 to 4500 grams.

Exclusion Criteria:

* Medical disorders and hypertensive disorders of pregnancy.
* Intrauterine fetal death.
* Known or suspected fetal anomalies.
* Oxytocin induction or augmented cases.
* Obstetrical complications (bleeding, premature rupture of membranes).
* Previous CS or Previous Myomectomy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women between 18-35 years of age with normal pregnancy
Enrollment: 150 (Estimated)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Duration of the third stage of labor. | 5-15 minutes
  Duration of placental expulsion from the uterus after delivery of the fetus. by the use of a stop watch to calculate the time in minutes and seconds passing starting from the delivery of the baby till delivery of the placenta outside the the vagina.
  To compare How long does the 3rd stage of labor persist with each intervention (in minutes and seconds).

SECONDARY OUTCOMES:
Retained placenta | >30 minutes
  defined as a placenta that remained in the uterus for 30 minutes or more after delivery.
  by the use of a stop watch to calculate the time in minutes and seconds needed for placental expulsion.
  To compare which intervention can result in delayed expulsion of placenta (in minutes and seconds) and cause a retained placenta.
the Need for manual removal of placenta | > 30 minutes
  manual removal of the placenta under general anesthesia if the placental expulsion is delayed for more than 30 minutes.
  to compare which intervention will require manual removal of the retained(by the percentage of yes and no) placenta.
the drop in hemoglobin in gm/dl | after 2 hours
  hemoglobin concentration in gm/dl will be measured for all participants before onset of delivery of the baby and 2 hours after labour and compare which maneuver included increased blood loss determined by the difference of hemoglobin concentration in gm/dl in the basal Hb level and the 2hr later Hb level.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer F Borg, MD, Study Director — Ain Shams University; Bassem I Ali, MD, Study Director — Ain Shams University; Islam M Abbas, MBBch, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol